CLINICAL TRIAL: NCT03306329
Title: A Phase 2a, Double-Blind, Placebo-Controlled Two-Part Study To Investigate the Safety and Efficacy of Increasing Doses Of DNS-7801 In Parkinson's Disease (PD) Subjects With Motor Fluctuations
Brief Title: DNS-7801 vs. Placebo in Parkinson's Disease
Acronym: PRIORITY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative
Sponsor: Dart NeuroScience, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNS-7801-201
Record Dates: First submitted 2017-09-25; First posted 2017-10-11 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DNS-7801 (low-dose) (Experimental)
  Interventions: Drug: DNS-7801 (low-dose)
- DNS-7801 (high-dose) (Experimental)
  Interventions: Drug: DNS-7801 (high dose)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNS-7801 (low-dose) — DNS-7801 (low-dose) tablets administered once daily.
  Arms: DNS-7801 (low-dose)
Drug: DNS-7801 (high dose) — DNS-7801 (high dose) tablets administered once daily.
  Arms: DNS-7801 (high-dose)
Drug: Placebo — Placebo tablets administered once daily
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, two-part placebo-controlled parallel group outpatient treatment study that will utilize standard Parkinson's Disease measures to evaluate the effect of DNS-7801

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects who are diagnosed with Parkinson's disease as defined by the United Kingdom PD Society Brain Bank Criteria for the Diagnosis of PD.
* Modified Hoehn and Yahr Staging ≤ 3 in ON state.
* Mini Mental State Examination Score ≥ 26.
* Subjects must currently have a good response to levodopa and be receiving a stable dose of levodopa ( at least 4 doses per day of standard levodopa or ≥ 3 doses per day of Rytary™ (Carbidopa and levodopa Extended-Release Capsules) for at least 4 weeks prior to screening).
* Subjects must experience motor fluctuations with at least 2 hours of OFF periods each day in the awake time.
* Subjects must experience predictable early morning OFF periods.
* Subjects must be able to come to the clinic in the practically defined OFF state.
* Subject must have achieved the following results for home PD diary training, practice diary collection, and Baseline diary recordings (PART B ONLY):

  * During a diary concordance session with an approved PD diary trainer/rater (minimum 4 hours), subject achieved at least 80% overall diary concordance, including at least 1 OFF interval.
  * Returned a valid 2-day (i.e., 2 consecutive 24-hour periods) practice home PD diary (as defined below).
  * Returned valid diary recordings preceding the Baseline Visit that indicated at least 2 hours of OFF time on each of the 2 days.
* All anti-parkinsonian medications must be maintained at a stable dose for at least 4 weeks prior to the initial Screening Visit with the exception of monoamine oxidase-B inhibitors, which must be maintained at a stable level for at least 8 weeks prior to the screening visit.

Main Exclusion Criteria:

* Diagnosis of secondary or an atypical Parkinsonian syndrome.
* Subject has severe disabling dyskinesia.
* Subject has clinically significant psychosis or hallucinations or history of psychosis in past 6 months.
* History of previous neurosurgery for PD.
* Currently or previously on Duopa/Duodopa.
* Currently on apomorphine or have received apomorphine within 30 days prior to baseline.
* The subject has a diagnosis or history of a substance related disorder (excluding nicotine and caffeine), including alcohol related disorder (Diagnostic and Statistical Manual of Mental Disorders 5 criteria) during the 12 months prior to the Screening Visit.
* The subject has tested positive at the Screening Visit for drugs of abuse (e.g., opiates, cannabinoids, methadone, cocaine, and amphetamines [including ecstasy]).
* Any medical (including acute or chronic pain), surgical, or psychiatric condition, laboratory value, or concomitant medication which, in the opinion of the Investigator or the eligibility reviewer, makes the subject unsuitable for study entry or potentially unable to complete all aspects of the study.
* Suicidal ideation within 1 year prior to the Screening Visit as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the Columbia Suicide Severity Rating Scale (C-SSRS) or attempted suicide within the last 5 years.
* Subjects with a current major depressive episode or a Beck Depression Inventory-II score of > 19. Subjects receiving treatment for depression with antidepressants may be enrolled if they have been on a stable daily dose of the antidepressant for at least 8 weeks before the Baseline Visit.
* Exposure to neuroleptics (antipsychotic drugs) for more than 1 month within the past 2 years, or any exposure within the past year.
* Any malignancy in the 5 years prior to randomization (excluding basal cell carcinoma of the skin or cervical carcinoma in situ that have been successfully treated).
* Current or previous diagnosis of malignant melanoma or the presence of any suspicious skin lesion based on physical exam findings.
* Subjects, who, for any reason, are judged by the Investigator to be inappropriate for this study, including subjects who are unable to communicate or cooperate with the Investigator or who have/had a clinically significant illness or abnormal physical examination that may compromise safety of the subject during the trial or affect ability of the subject to adhere to study procedures
* Serum creatinine > 2 mg/dL.
* Total serum bilirubin > 2 mg/dL.
* Coagulation parameters (prothrombin time, activated partial thromboplastin time and international normalized ratio) and other laboratory parameters that, in the opinion of the Investigator, are in a range that could be harmful to the subject.
* Subjects with alanine transaminase or aspartate transaminase ≥ 3x upper limit of normal at Screening.
* Uncontrolled hypertension (e.g., Stage 2 hypertension - systolic > 160 mm Hg or diastolic > 100 mm Hg).
* Orthostatic hypotension that is symptomatic or requires medication.
* Subjects with heart block that, in the opinion of the Investigator, could interfere with the subject's ability to participate in the study.
* Hospitalization for myocardial infarction, ischemic heart disease, or congestive heart failure within the 12 months prior to the Screening Visit.
* Evidence on clinical examination or ECG of a clinically significant arrhythmia, as assessed by the Investigator.
* Subject is currently lactating or pregnant or planning to become pregnant during the study.
* Use of any medications that are prohibited concomitant medications during the study, are known to be strong or moderate inducers or inhibitors of cytochrome P450 (CYP) 3A4, or are contraindicated for treatment with study drug.
* Consumption of grapefruit containing foods or beverages within 14 days before Baseline and for 14 days after the last dose of study drug.
* Subject is currently participating in or has participated in another study of a study drug or medical device in the last 3 months or within 5 half-lives of the study drug (whichever is longer) prior to Baseline.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Part A: Maximal change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III from predose | 2-days
Part B: Change in OFF time from Baseline to Day 28 on home PD diary | 28-days

SECONDARY OUTCOMES:
Part A: Safety of DNS-7801 evaluating the number of Treatment Emergent Adverse Events (TEAEs) at each study visit | 17-days
Part A: Score on the Columbia Suicide Severity Rating Scale (C-SSRS) as assessed at each study visit | 17-days
Part A: Tolerability of DNS-7801 assessed by discontinuation due to TEAE(s) [percent completers] at Day 10 | 10-days
Part B: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III from Baseline to Day 28 | 28-days
Part B: Change in ON time without troublesome dyskinesia from Baseline to Day 28 | 28-days
Part B: Change from Baseline in the Parkinson's Disease Quality of Life Questionnaire Summary Index | 28-days
Part B: Proportion of subjects with improvement in Clinical Global Impression of Improvement (CGI-I) | 28-days
Part B: Safety of DNS-7801 evaluating the number of Treatment Emergent Adverse Events (TEAEs) at each study visit | 35-days
Part B: Score on the Columbia Suicide Severity Rating Scale (C-SSRS) as assessed at each study visit | 35-days
Part B: Tolerability of DNS-7801 assessed by discontinuation due to TEAE(s) [percent completers] | 28-days

CONTACTS AND LOCATIONS:
Overall Officials: Philip Perera, MD, Study Director — Dart NeuroScience, LLC
Locations (9):
- United States (9):
  - Collaborative Neuroscience Network, Long Beach, California
  - SC3 Research, Pasadena, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Parkinsons Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of South Florida Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Quest Research Institute, Farmington, Michigan
  - Washington University, St Louis, Missouri
  - The Neurological Institute PA, Charlotte, North Carolina
  - Premier Clinical Research, Spokane, Washington